CLINICAL TRIAL: NCT02001987
Title: A Multi-Center Open-Label Study to Evaluate the Efficacy, Safety and Tolerability of Subcutaneous Tocilizumab in Tocilizumab-Naive Patients With Active Rheumatoid Arthritis Who Have an Inadequate Response to Current Non-Biologic DMARD and/or Biologic Therapy
Brief Title: A Study of Tocilizumab (RoActemra) in Tocilizumab-Naive Participants With Rheumatoid Arthritis and Inadequate Response to Non-Biologic Disease-Modifying Antirheumatic Drugs (DMARDs) and/or Biologic Therapy
Acronym: TOSCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28693; 2013-001718-14 (EudraCT Number)
Record Dates: First submitted 2013-11-29; First posted 2013-12-05 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

ARMS (1):
- Tocilizumab (Experimental): Participants will receive tocilizumab at a dose of 162 milligrams (mg) as subcutaneous (SC) injection once a week administered as monotherapy or in combination with methotrexate or other csDMARDs (at investigator's discretion) for 24 weeks. Participants who complete the core study period will be allowed to enter a long-term-extension (LTE) period to continue study treatment for up to a maximum of another 52 weeks or until the commercial availability of SC tocilizumab, whichever occurs first.
  Interventions: Drug: Tocilizumab; Drug: Methotrexate; Drug: csDMARDs

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab will be administered at a dose of 162 mg as SC injection once a week.
  Other Names: RoActemra; RO4877533
Drug: Methotrexate — Methotrexate will be administered at a stable dose that was initiated at least 4 weeks prior to Baseline, at investigator's discretion.
Drug: csDMARDs — csDMARDs (at investigator's discretion) will be administered at a stable dose that was initiated at least 4 weeks prior to Baseline, at investigator's discretion.

SUMMARY:
This two part, multi-center, open-label, single-arm study will evaluate the efficacy and safety of tocilizumab as a monotherapy or in combination with methotrexate or other conventional synthetic disease modifying antirheumatic drugs (csDMARDs) in participants with moderate to severe active rheumatoid arthritis who have an inadequate response or are intolerant to non-biologic csDMARDs and/or biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of active rheumatoid arthritis according to the revised (1987) ACR criteria or EULAR/ACR (2010) criteria and receiving outpatient treatment
* Oral corticosteroids (</= 10 mg/day prednisone or equivalent), nonsteroidal anti-inflammatory drugs (NSAIDs), and permitted csDMARDs are allowed at a stable dose for at least 4 weeks prior to Baseline
* At Screening either CRP >/=10 mg/L or ESR >/=20 mm/h and SJC >/=3 (based on 44 joints)
* Inadequate response (IR) to tumor necrosis factor, abatacept and/or non-biological DMARDs

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to Screening or planned major surgery within 6 months following Baseline
* Rheumatic autoimmune disease other than rheumatoid arthritis; Secondary Sjögren's syndrome with rheumatoid arthritis is permitted
* Functional Class IV as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Diagnosis of juvenile idiopathic arthritis or juvenile rheumatoid arthritis and/or rheumatoid arthritis before the age of 16
* Prior history of or current inflammatory joint disease other than rheumatoid arthritis
* Exposure to tocilizumab at any time prior to Baseline
* Treatment with any investigational agent within 4 weeks (or five half-lives of the investigational drug, whichever was longer) of Screening
* Previous treatment with any cell-depleting therapies, including investigational agents or approved therapies or any alkylating agents such as chlorambucil, or with total lymphoid irradiation
* Treatment with IV gamma globulin, plasmapheresis within 6 months of Baseline
* Intraarticular or parenteral corticosteroids within 4 weeks prior to Baseline
* Immunization with a live/attenuated vaccine within 4 weeks prior to Baseline
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Serious uncontrolled concomitant disease or other significant condition
* History of diverticulitis, diverticulosis requiring antibiotic treatment, or chronic ulcerative lower gastrointestinal disease
* Current or history of recurrent bacterial, viral, fungal, mycobacterial, or other infections
* Any infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of Screening or oral antibiotics within 2 weeks of Screening
* Active tuberculosis requiring treatment within the previous 3 years
* Positive for hepatitis B or C
* Primary or secondary immunodeficiency disorder
* Active cancer, or cancer diagnosed within the previous 10 years (except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised or cured), or breast cancer diagnosed within the previous 20 years
* History of alcohol, drug, or chemical abuse within 1 year prior to Screening
* Neuropathies or other conditions that might interfere with pain evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- France (27):
  - Amiens
  - Bordeaux
  - Brest
  - Caen
  - Cahors
  - Clermont-Ferrand
  - Échirolles
  - La Source
  - Le Mans
  - Lille
  - Limoges
  - Lomme
  - Lyon
  - Marseille
  - Metz-Tessy
  - Monaco
  - Montpellier
  - Mulhouse
  - Paris
  - Rennes
  - Rouen
  - Saint-Mandé
  - Saint-Priest-en-Jarez
  - Strasbourg
  - Thonon-les-Bains
  - Toulouse
  - Vandœuvre-lès-Nancy

REFERENCES:
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Devenport J, Petho-Schramm A. Effects of concomitant glucocorticoids in TOZURA, a common-framework study programme of subcutaneous tocilizumab in rheumatoid arthritis. Rheumatology (Oxford). 2019 Jun 1;58(6):1056-1064. doi: 10.1093/rheumatology/key393. PMID 30649524
- [Derived] Choy E, Caporali R, Xavier R, Fautrel B, Sanmarti R, Bao M, Bernasconi C, Petho-Schramm A. Subcutaneous tocilizumab in rheumatoid arthritis: findings from the common-framework phase 4 study programme TOZURA conducted in 22 countries. Rheumatology (Oxford). 2018 Mar 1;57(3):499-507. doi: 10.1093/rheumatology/kex443. PMID 29244149

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 183 participants were screened; 139 participants were eligible for the study and assigned to study treatment.
Pre-assignment Details: Analyses of primary/ secondary outcome measures were planned and performed in different analysis populations described in respective analysis population descriptions. Analyses of few secondary outcome measures and adverse events were planned and performed according to predefined subgroup populations and have been presented accordingly.
Groups:
- TCZ - All Participants: Participants in core study period received tocilizumab (TCZ, RoActemra) at a dose of 162 milligrams (mg) as subcutaneous (SC) injection once a week as monotherapy or in combination with Methotrexate (MTX) or other Conventional Synthetic Disease-Modifying Antirheumatic Drugs (csDMARDs) (at investigator's discretion) for 24 weeks. Participants who completed the core study period were allowed to enter a Long-term-extension (LTE) period to continue study treatment for up to a maximum of another 52 weeks or until the commercial availability of SC TCZ, whichever came first.
Period: Core Study Period (24 Weeks)
Arm/Group | TCZ - All Participants
Started | 139
Completed | 116
Not Completed | 23
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Non-Serious Hypersensitivity Reaction | 2
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 3
Not completed — Lack of Efficacy | 3
Period: LTE Period (52 Weeks)
Arm/Group | TCZ - All Participants
Started | 116
Completed | 107
Not Completed | 9
Not completed — Lost to Follow-up | 2
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lack of Efficacy | 1
Not completed — Other | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who received at least one dose of SC TCZ.
Groups:
- TCZ - All Participants: Participants in core study period received TCZ at a dose of 162 mg as SC injection once a week as monotherapy or in combination with MTX or other csDMARDs (at investigator's discretion) for 24 weeks. Participants who completed the core study period were allowed to enter a LTE period to continue study treatment for up to a maximum of another 52 weeks or until the commercial availability of SC TCZ, whichever came first.
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 36

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Disease Activity Score Based on 28-joints Count and Erythrocyte Sedimentation Rate (DAS28-ESR) at Week 24
Description: The DAS28-ESR was derived from assessments of erythrocyte sedimentation rate (ESR), tender joint count (TJC), swollen joint count (SJC), and Patient Global Assessment of disease activity (PGA) according to 100-millimeter (mm) Visual Analog Scale (VAS). DAS28-ESR scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of painful joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in millimeters per hour (mm/h). DAS28-ESR scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to Week 24 was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline, Week 24
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure. In case of missing value, Last Observation Carried Forward (LOCF) method was applied.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- TCZ - All Participants - Core Study Period: Participants in core study period received TCZ at a dose of 162 mg as SC injection once a week as monotherapy or in combination with MTX or other csDMARDs (at investigator's discretion) for 24 weeks.
Arm/Group | TCZ - All Participants - Core Study Period
Number analyzed (Participants) | 136
units on a scale
  Baseline | 5.80 (1.14)
  Change at Week 24 | -3.07 (1.52)

2. Secondary Outcome: Change From Baseline in DAS28-ESR at Weeks 2, 4, 8, 12, 16, 20, and 24
Description: The DAS28-ESR was derived from assessments of ESR, TJC, SJC, and PGA according to 100-mm VAS. DAS28-ESR scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of painful joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28-ESR scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to any time point was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable at specified time points for different arms, respectively. In case of missing value at Week 24, LOCF method was applied.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- TCZ MONO - Core Study Period: Participants who did not receive treatment with any csDMARDs 4 weeks prior first TCZ administration and received monotherapy with TCZ at a dose of 162 mg as SC injection once a week for 24 weeks.
- TCZ COMBO - Core Study Period: Participants who received treatment with MTX or other csDMARDs 4 weeks prior first TCZ administration and/or received TCZ at a dose of 162 mg as SC injection once a week in combination with MTX or other csDMARDs (at investigator's discretion) for 24 weeks.
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 42 | 94
units on a scale
  Baseline | 6.08 (1.21) | 5.67 (1.10)
  Change at Week 2: number analyzed (Participants) | 40 | 87
  Change at Week 2 | -1.19 (1.05) | -1.41 (1.03)
  Change at Week 4: number analyzed (Participants) | 37 | 88
  Change at Week 4 | -2.16 (1.17) | -2.21 (1.14)
  Change at Week 8: number analyzed (Participants) | 37 | 87
  Change at Week 8 | -2.70 (1.40) | -2.74 (1.36)
  Change at Week 12: number analyzed (Participants) | 36 | 82
  Change at Week 12 | -3.16 (1.54) | -3.02 (1.33)
  Change at Week 16: number analyzed (Participants) | 34 | 81
  Change at Week 16 | -3.20 (1.59) | -3.08 (1.29)
  Change at Week 20: number analyzed (Participants) | 33 | 77
  Change at Week 20 | -3.27 (1.35) | -3.21 (1.43)
  Change at Week 24 | -3.01 (1.62) | -3.10 (1.48)

3. Secondary Outcome: Percentage of Participants With DAS28-ESR Low Disease Activity (LDA) and Remission at Week 24
Description: The DAS28-ESR was derived from assessments of ESR, TJC, SJC, and PGA according to 100-mm VAS. DAS28-ESR scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of painful joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28-ESR scores could range from 0 to 10, where higher scores represented higher disease activity. DAS28-ESR score less than or equal to (</=) 3.2 indicates LDA, DAS28-ESR score greater than (>) 3.2 indicates moderate to high disease activity, and DAS28-ESR less than (<) 2.6 indicates remission. Percentage of participants with DAS28-ESR LDA and remission at Week 24 is reported. 95 percent (%) confidence interval (CI) was determined using Clopper-Pearson method.
Time Frame: Week 24
Population: FAS; In case of missing value at Week 24, LOCF method was applied.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 43 | 96
percentage of participants
  LDA | 67.4 [51.46 to 80.92] | 70.8 [60.67 to 79.67]
  Remission | 41.9 [27.01 to 57.87] | 55.2 [44.71 to 65.37]

4. Secondary Outcome: Change From Baseline in DAS28-ESR at Week 24 and at Last Assessment
Description: The DAS28-ESR was derived from assessments of ESR, TJC, SJC, and PGA according to 100-millimeter (mm) VAS. DAS28-ESR scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of painful joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28-ESR scores could range from 0 to 10, where higher scores represented higher disease activity. The change from Baseline to any time point was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline, Week 24, last assessment (up to Week 76)
Population: LTE population included all FAS participants who received at least one dose of SC TCZ after Week 24 visit. Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure. In case of missing value at Week 24, LOCF method was applied.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 63
units on a scale
  Baseline | 5.90 (1.26)
  Change at Week 24 | -3.30 (1.44)
  Change at Last Assessment | -3.41 (1.47)

5. Secondary Outcome: Percentage of Participants With DAS28-ESR LDA and Remission at Week 24 and at Last Assessment
Description: The DAS28-ESR was derived from assessments of ESR, TJC, SJC, and PGA according to 100-mm VAS. DAS28-ESR scores were calculated as [0.56 × square root of TJC] + [0.28 × square root of SJC] + [0.70 × natural log (ESR)] + [0.014 × VAS]. TJC was defined as the number of painful joints and SJC was defined as the number of swollen joints, each assessed on 28 joints. ESR was measured in mm/h. DAS28-ESR scores could range from 0 to 10, where higher scores represented higher disease activity. DAS28-ESR score </=3.2 indicates LDA, DAS28-ESR score >3.2 indicates moderate to high disease activity, and DAS28-ESR <2.6 indicates remission. Percentage of participants with DAS28-ESR LDA and remission at Week 24 and at last assessment is reported.
Time Frame: Week 24, last assessment (up to Week 76)
Population: LTE population; In case of missing value at Week 24, LOCF method was applied.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 64
percentage of participants
  Week 24, LDA | 71.9
  Week 24, Remission | 54.7
  Last Assessment, LDA | 71.9
  Last Assessment, Remission | 53.1

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20% (ACR20), 50% (ACR50), and 70% (ACR70) Response at Week 24
Description: The ACR 20, 50, and 70 responses at any time was defined as greater than or equal to (>/=) 20%, 50%, and 70% improvement compared to baseline in TJC (assessed on 68 joints) and SJC (assessed on 66 joints); and 20%, 50%, 70% improvement compared to baseline in 3 of the following 5 criteria, respectively: 1) PGA according to 100-mm VAS, 2) Physician's global assessment of disease activity according to 100-mm VAS, 3) participant's global assessment of pain according to 100-mm VAS, 4) Participant's assessment of functional ability via a Health Assessment Questionnaire-Disability Index (HAQ-DI), and 5) Acute phase reactant (ESR in mm/h or C-Reactive Protein [CRP] in milligrams per liter [mg/L]). Percentage of participants with ACR 20, 50, and 70 responses at Week 24 is reported. 95% CI was determined using Clopper-Pearson method.
Time Frame: Baseline, Week 24
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure. Missing data was considered as non-response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 33 | 84
percentage of participants
  ACR20 | 69.7 [51.29 to 84.41] | 73.8 [63.07 to 82.80]
  ACR50 | 54.5 [36.35 to 71.89] | 52.4 [41.19 to 63.40]
  ACR70 | 33.3 [17.96 to 51.83] | 28.6 [19.24 to 39.47]

7. Secondary Outcome: Percentage of Participants Achieving ACR20, ACR50, and ACR70 Response at Week 24 and at Last Assessment
Description: The ACR 20, 50, and 70 responses at any time is defined as >/=20%, 50%, and 70% improvement compared to baseline in TJC (assessed on 68 joints) and SJC (assessed on 66 joints); and 20%, 50%, 70% improvement compared to baseline in 3 of the following 5 criteria, respectively: 1) PGA according to 100-mm VAS, 2) Physician's global assessment of disease activity according to 100-mm VAS, 3) participant's global assessment of pain according to 100-mm VAS, 4) Participant's assessment of functional ability via HAQ-DI, and 5) Acute phase reactant (ESR in mm/h or CRP in mg/L). Percentage of participants with ACR 20, 50, and 70 responses at Week 24 and at last assessment is reported.
Time Frame: Baseline, Week 24, last assessment (up to Week 76)
Population: LTE population; Missing data was considered as non-response.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 64
percentage of participants
  Week 24, ACR20 | 76.6
  Week 24, ACR50 | 51.6
  Week 24, ACR70 | 35.9
  Last Assessment, ACR20 | 76.6
  Last Assessment, ACR50 | 56.3
  Last Assessment, ACR70 | 37.5

8. Secondary Outcome: Percentage of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28-ESR at Week 24
Description: The DAS28-ESR-based EULAR response criteria were used to measure individual response as 'Good', 'Moderate', and 'No Response', depending upon DAS28-ESR absolute scores at Week 24 and the DAS28-ESR reduction from Baseline to Week 24. Good Response: change from baseline >1.2 with DAS28-ESR score </=3.2; Moderate Response: change from baseline >1.2 with DAS28-ESR score >3.2 to </=5.1 or change from baseline >0.6 to </=1.2 with DAS28-ESR score </=5.1; No Response: change from baseline </=0.6 or change from baseline >0.6 and </=1.2 with DAS28-ESR score >5.1. Percentage of participants with EULAR responses at Week 24 is reported. 95% CI was determined using Clopper-Pearson method.
Time Frame: Baseline, Week 24
Population: FAS; Missing data was considered as non-response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 43 | 96
percentage of participants
  Good Response | 58.1 [42.13 to 72.99] | 60.4 [49.92 to 70.25]
  Moderate Response | 14.0 [5.30 to 27.93] | 19.8 [12.36 to 29.17]
  No Response | 27.9 [15.33 to 43.67] | 19.8 [12.36 to 29.17]

9. Secondary Outcome: Percentage of Participants With EULAR Response Based on DAS28-ESR at Week 24 and at Last Assessment
Description: The DAS28-ESR-based EULAR response criteria were used to measure individual response as 'Good', 'Moderate', and 'No Response', depending upon DAS28-ESR absolute scores at Week 24 and the DAS28-ESR reduction from Baseline to Week 24. Good Response: change from baseline >1.2 with DAS28-ESR score </=3.2; Moderate Response: change from baseline >1.2 with DAS28-ESR score >3.2 to </=5.1 or change from baseline >0.6 to </=1.2 with DAS28-ESR score </=5.1; No Response: change from baseline </=0.6 or change from baseline >0.6 and </=1.2 with DAS28-ESR score >5.1. Percentage of participants with EULAR responses at Week 24 and at last assessment is reported.
Time Frame: Baseline, Week 24, last assessment (up to Week 76)
Population: LTE population; Missing data was considered as non-response.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 64
percentage of participants
  Week 24, Good Response | 68.8
  Week 24, Moderate Response | 26.6
  Week 24, No Response | 4.7
  Last Assessment, Good Response | 65.6
  Last Assessment, Moderate Response | 31.3
  Last Assessment, No Response | 3.1

10. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 2, 4, 8, 12, 16, 20, and 24
Description: SDAI is a numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and Physician's global assessment of disease activity according to 100-mm VAS and CRP in mg per deciliter (dL). Higher scores indicate greater affection due to disease activity. SDAI total score = 0-86. SDAI </=3.3 indicates disease remission, </=11 indicates LDA, </=26 indicates moderate disease activity, and >26 indicates high disease activity. The change from Baseline to any time point was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 39 | 90
units on a scale
  Baseline | 35.42 (12.61) | 31.47 (11.77)
  Change at Week 2: number analyzed (Participants) | 38 | 84
  Change at Week 2 | -8.54 (10.67) | -9.20 (9.37)
  Change at Week 4: number analyzed (Participants) | 37 | 83
  Change at Week 4 | -14.23 (10.76) | -14.62 (11.33)
  Change at Week 8: number analyzed (Participants) | 35 | 82
  Change at Week 8 | -20.20 (13.22) | -17.47 (12.47)
  Change at Week 12: number analyzed (Participants) | 34 | 79
  Change at Week 12 | -23.09 (13.82) | -20.33 (12.97)
  Change at Week 16: number analyzed (Participants) | 29 | 76
  Change at Week 16 | -24.31 (15.14) | -21.39 (12.66)
  Change at Week 20: number analyzed (Participants) | 29 | 71
  Change at Week 20 | -24.41 (15.28) | -21.93 (13.35)
  Change at Week 24 | -22.45 (14.48) | -20.31 (13.34)

11. Secondary Outcome: Percentage of Participants With SDAI LDA and Remission at Week 24
Description: SDAI is a numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and Physician's global assessment of disease activity according to 100-mm VAS and CRP in mg/dL. Higher scores indicate greater affection due to disease activity. SDAI total score = 0-86. SDAI </=3.3 indicates disease remission, </=11 indicates LDA, </=26 indicates moderate disease activity, and >26 indicates high disease activity. Percentage of participants with SDAI LDA and remission at Week 24 is reported. 95% CI was determined using Clopper-Pearson method.
Time Frame: Week 24
Population: FAS; Missing data was considered as non-response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 43 | 96
percentage of participants
  LDA | 46.5 [31.18 to 62.35] | 59.4 [48.87 to 69.29]
  Remission | 18.6 [8.39 to 33.40] | 19.8 [12.36 to 29.17]

12. Secondary Outcome: Change From Baseline in SDAI at Week 24 and at Last Assessment
Description: SDAI is a numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and Physician's global assessment of disease activity according to 100-mm VAS and CRP in mg/dL. Higher scores indicate greater affection due to disease activity. SDAI total score = 0-86. SDAI </=3.3 indicates disease remission, </=11 indicates LDA, </=26 indicates moderate disease activity, and >26 indicates high disease activity. The change from Baseline to any time point was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline, Week 24, last assessment (up to Week 76)
Population: LTE population; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable at specified time points. In case of missing value at Week 24, LOCF method was applied.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 57
units on a scale
  Change at Week 24 | -23.29 (13.81)
  Change at Last Assessment: number analyzed (Participants) | 55
  Change at Last Assessment | -24.36 (12.61)

13. Secondary Outcome: Percentage of Participants With SDAI LDA and Remission at Week 24 and at Last Assessment
Description: SDAI is a numerical sum of 5 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and Physician's global assessment of disease activity according to 100-mm VAS and CRP in mg/dL. Higher scores indicate greater affection due to disease activity. SDAI total score = 0-86. SDAI </=3.3 indicates disease remission, </=11 indicates LDA, </=26 indicates moderate disease activity, and >26 indicates high disease activity. Percentage of participants with SDAI LDA and remission at Week 24 and at last assessment is reported.
Time Frame: Week 24, last assessment (up to Week 76)
Population: LTE population; Missing data was considered as non-response.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 64
percentage of participants
  Week 24, LDA | 57.8
  Week 24, Remission | 20.3
  Last Assessment, LDA | 64.1
  Last Assessment, Remission | 25.0

14. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 2, 4, 8, 12, 16, 20, and 24
Description: CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and Physician's global assessment of disease activity according to 100-mm VAS. Higher scores represent greater affection due to disease activity. CDAI total score = 0-76. CDAI score </=2.8 indicates disease remission, </=10 indicates LDA, </=22 indicates moderate disease activity, and >22 indicates high disease activity. The change from Baseline to any time point was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 39 | 90
units on a scale
  Baseline | 32.17 (11.11) | 29.34 (11.05)
  Change at Week 2: number analyzed (Participants) | 38 | 84
  Change at Week 2 | -5.57 (9.69) | -7.15 (8.87)
  Change at Week 4: number analyzed (Participants) | 37 | 85
  Change at Week 4 | -11.17 (10.14) | -12.65 (10.97)
  Change at Week 8: number analyzed (Participants) | 35 | 85
  Change at Week 8 | -17.32 (12.00) | -15.75 (11.62)
  Change at Week 12: number analyzed (Participants) | 34 | 79
  Change at Week 12 | -20.25 (12.50) | -18.17 (12.20)
  Change at Week 16: number analyzed (Participants) | 32 | 77
  Change at Week 16 | -20.24 (14.13) | -19.25 (11.88)
  Change at Week 20: number analyzed (Participants) | 30 | 74
  Change at Week 20 | -21.27 (13.58) | -19.29 (12.82)
  Change at Week 24 | -19.45 (13.34) | -18.40 (12.78)

15. Secondary Outcome: Percentage of Participants With CDAI LDA and Remission at Week 24
Description: CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and Physician's global assessment of disease activity according to 100-mm VAS. Higher scores represent greater affection due to disease activity. CDAI total score = 0-76. CDAI score </=2.8 indicates disease remission, </=10 indicates LDA, </=22 indicates moderate disease activity, and >22 indicates high disease activity. Percentage of participants with CDAI LDA and remission at Week 24 is reported. 95% CI was determined using Clopper-Pearson method.
Time Frame: Week 24
Population: FAS; Missing data was considered as non-response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 43 | 96
percentage of participants
  LDA | 44.2 [29.08 to 60.12] | 60.4 [49.92 to 70.25]
  Remission | 16.3 [6.81 to 30.70] | 16.7 [9.84 to 25.65]

16. Secondary Outcome: Change From Baseline in CDAI at Week 24 and at Last Assessment
Description: as for outcome 14
Time Frame: Baseline, Week 24, last assessment (up to Week 76)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 57
units on a scale
  Change at Week 24 | -20.85 (13.06)
  Change at Last Assessment: number analyzed (Participants) | 55
  Change at Last Assessment | -21.74 (12.06)

17. Secondary Outcome: Percentage of Participants With CDAI LDA and Remission at Week 24 and at Last Assessment
Description: CDAI is a numerical sum of 4 outcome parameters: TJC and SJC based on a 28-joint assessment, PGA and Physician's global assessment of disease activity according to 100-mm VAS. Higher scores represent greater affection due to disease activity. CDAI total score = 0-76. CDAI score </=2.8 indicates disease remission, </=10 indicates LDA, </=22 indicates moderate disease activity, and >22 indicates high disease activity. Percentage of participants with CDAI LDA and remission at Week 24 and at last assessment is reported.
Time Frame: Week 24, last assessment (up to Week 76)
Population: LTE population; Missing data was considered as non-response.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 64
percentage of participants
  Week 24, LDA | 57.8
  Week 24, Remission | 17.2
  Last Assessment, LDA | 60.9
  Last Assessment, Remission | 23.4

18. Secondary Outcome: Change From Baseline in SJC at Weeks 2, 4, 8, 12, 16, 20, and 24
Description: A total of 28 joints were assessed for swelling. The number of swollen joints at could range from 0 to 28, where higher values represented more swollen joints. The change from Baseline to any time point was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: FAS; Here, 'Number Analyzed' signifies number of participants evaluable at specified time points for different arms, respectively. In case of missing value at Week 24, LOCF method was applied.
Measure: Median (Full Range); unit: swollen joints
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 43 | 96
swollen joints
  Baseline | 6.0 [0.0 to 24.0] | 7.0 [0.0 to 23.0]
  Change at Week 2: number analyzed (Participants) | 42 | 95
  Change at Week 2 | -1.0 [-9.0 to 14.0] | -2.0 [-13.0 to 8.0]
  Change at Week 4: number analyzed (Participants) | 40 | 94
  Change at Week 4 | -3.0 [-8.0 to 4.0] | -3.0 [-18.0 to 5.0]
  Change at Week 8: number analyzed (Participants) | 38 | 92
  Change at Week 8 | -3.5 [-18.0 to 6.0] | -4.0 [-17.0 to 3.0]
  Change at Week 12: number analyzed (Participants) | 37 | 89
  Change at Week 12 | -4.0 [-22.0 to 3.0] | -5.0 [-23.0 to 2.0]
  Change at Week 16: number analyzed (Participants) | 35 | 88
  Change at Week 16 | -5.0 [-22.0 to 6.0] | -5.0 [-23.0 to 2.0]
  Change at Week 20: number analyzed (Participants) | 35 | 84
  Change at Week 20 | -4.0 [-21.0 to 3.0] | -5.0 [-22.0 to 4.0]
  Change at Week 24 | -5.0 [-21.0 to 14.0] | -5.0 [-23.0 to 2.0]

19. Secondary Outcome: Change From Baseline in SJC at Week 24 and at Last Assessment
Description: as for outcome 18
Time Frame: Baseline, Week 24, last assessment (up to Week 76)
Population: LTE population; In case of missing value at Week 24, LOCF method was applied.
Measure: Median (Full Range); unit: swollen joints
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 64
swollen joints
  Change at Week 24 | -6.0 [-23.0 to 2.0]
  Change at Last Assessment | -6.5 [-22.0 to 5.0]

20. Secondary Outcome: Change From Baseline in TJC at Weeks 2, 4, 8, 12, 16, 20, and 24
Description: A total of 28 joints were assessed for tenderness. The number of tender joints at could range from 0 to 28, where higher values represented more tender joints. The change from Baseline to any time points was averaged among all participants, where negative changes indicated an improvement in disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: as for outcome 18
Measure: Median (Full Range); unit: tender joints
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 43 | 96
tender joints
  Baseline | 12.0 [0.0 to 28.0] | 8.0 [0.0 to 27.0]
  Change at Week 2: number analyzed (Participants) | 42 | 95
  Change at Week 2 | -1.0 [-13.0 to 12.0] | -2.0 [-18.0 to 12.0]
  Change at Week 4: number analyzed (Participants) | 40 | 94
  Change at Week 4 | -2.5 [-17.0 to 4.0] | -3.0 [-20.0 to 10.0]
  Change at Week 8: number analyzed (Participants) | 38 | 92
  Change at Week 8 | -6.5 [-19.0 to 12.0] | -5.0 [-21.0 to 8.0]
  Change at Week 12: number analyzed (Participants) | 37 | 89
  Change at Week 12 | -8.0 [-23.0 to 3.0] | -5.0 [-20.0 to 17.0]
  Change at Week 16: number analyzed (Participants) | 35 | 88
  Change at Week 16 | -8.0 [-24.0 to 8.0] | -5.5 [-23.0 to 4.0]
  Change at Week 20: number analyzed (Participants) | 35 | 84
  Change at Week 20 | -8.0 [-27.0 to 5.0] | -5.0 [-25.0 to 12.0]
  Change at Week 24 | -8.0 [-27.0 to 12.0] | -5.0 [-27.0 to 15.0]

21. Secondary Outcome: Change From Baseline in TJC at Week 24 and at Last Assessment
Description: as for outcome 20
Time Frame: Baseline, Week 24, last assessment (up to Week 76)
Population: LTE population; In case of missing value at Week 24, LOCF method was applied.
Measure: Median (Full Range); unit: tender joints
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 64
tender joints
  Change at Week 24 | -6.5 [-27.0 to 15.0]
  Change at Last Assessment | -6.0 [-27.0 to 9.0]

22. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Disease Activity at Weeks 2, 4, 8, 12, 16, 20, and 24
Description: Physician-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the physician's evaluation of disease activity (0 mm=none; 100 mm=very severe). The change from Baseline to any time point was averaged among all participants, where negative change indicated a decrease in physician-assessed disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, and 24
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable at specified time points. In case of missing value at Week 24, LOCF method was applied.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 132
mm
  Baseline | 62.08 (17.68)
  Change at Week 2: number analyzed (Participants) | 127
  Change at Week 2 | -11.38 (15.91)
  Change at Week 4: number analyzed (Participants) | 126
  Change at Week 4 | -22.10 (20.25)
  Change at Week 8: number analyzed (Participants) | 123
  Change at Week 8 | -29.67 (23.33)
  Change at Week 12: number analyzed (Participants) | 117
  Change at Week 12 | -35.25 (22.03)
  Change at Week 16: number analyzed (Participants) | 116
  Change at Week 16 | -35.69 (23.33)
  Change at Week 20: number analyzed (Participants) | 110
  Change at Week 20 | -37.80 (21.80)
  Change at Week 24 | -34.98 (22.43)

23. Secondary Outcome: Change From Baseline in PGA at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Description: Participant-assessed disease activity was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of disease activity (0 mm=none; 100 mm=very severe). The change from Baseline to any time point was averaged among all participants, where negative change indicated a decrease in participant-assessed disease activity.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: Quality of Life (QoL) population included all enrolled participants with at least one electronic patient-reported outcome (ePRO) questionnaire completed. Here, 'Overall Number of Participants Analyzed' = number of participants evaluable for this outcome measure and 'Number Analyzed' = number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 136
mm
  Baseline | 59.88 (24.14)
  Change at Week 2: number analyzed (Participants) | 131
  Change at Week 2 | -8.11 (21.64)
  Change at Week 4: number analyzed (Participants) | 130
  Change at Week 4 | -17.19 (25.71)
  Change at Week 8: number analyzed (Participants) | 127
  Change at Week 8 | -24.49 (29.94)
  Change at Week 12: number analyzed (Participants) | 121
  Change at Week 12 | -29.62 (29.84)
  Change at Week 16: number analyzed (Participants) | 115
  Change at Week 16 | -31.61 (28.89)
  Change at Week 20: number analyzed (Participants) | 112
  Change at Week 20 | -31.80 (31.16)
  Change at Week 24: number analyzed (Participants) | 113
  Change at Week 24 | -33.79 (31.19)
  Change at Week 28: number analyzed (Participants) | 60
  Change at Week 28 | -37.90 (29.87)
  Change at Week 32: number analyzed (Participants) | 51
  Change at Week 32 | -33.96 (32.19)
  Change at Week 36: number analyzed (Participants) | 39
  Change at Week 36 | -34.10 (30.05)
  Change at Week 40: number analyzed (Participants) | 23
  Change at Week 40 | -37.74 (28.63)
  Change at Week 44: number analyzed (Participants) | 20
  Change at Week 44 | -36.55 (26.27)
  Change at Week 48: number analyzed (Participants) | 16
  Change at Week 48 | -37.63 (26.07)
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -37.50 (33.25)
  Change at Week 56: number analyzed (Participants) | 6
  Change at Week 56 | -41.00 (41.91)
  Change at Week 60: number analyzed (Participants) | 2
  Change at Week 60 | -46.00 (49.50)
  Change at Week 64: number analyzed (Participants) | 2
  Change at Week 64 | -42.50 (53.03)

24. Secondary Outcome: Change From Baseline in Pain VAS Score at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Description: Participant-assessed pain was scored on a 100-mm VAS, where the distance from 0 mm represented the participant's self evaluation of pain (0 mm=none; 100 mm=very severe). The change from Baseline to any time point was averaged among all participants, where negative change indicated a decrease in participant-assessed pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: QoL population; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 135
mm
  Baseline | 57.57 (26.78)
  Change at Week 2: number analyzed (Participants) | 127
  Change at Week 2 | -7.50 (22.78)
  Change at Week 4: number analyzed (Participants) | 128
  Change at Week 4 | -15.28 (29.76)
  Change at Week 8: number analyzed (Participants) | 125
  Change at Week 8 | -22.58 (32.15)
  Change at Week 12: number analyzed (Participants) | 116
  Change at Week 12 | -28.29 (32.04)
  Change at Week 16: number analyzed (Participants) | 111
  Change at Week 16 | -29.50 (29.98)
  Change at Week 20: number analyzed (Participants) | 111
  Change at Week 20 | -30.55 (29.98)
  Change at Week 24: number analyzed (Participants) | 107
  Change at Week 24 | -31.85 (30.21)
  Change at Week 28: number analyzed (Participants) | 58
  Change at Week 28 | -33.29 (31.84)
  Change at Week 32: number analyzed (Participants) | 52
  Change at Week 32 | -32.67 (30.98)
  Change at Week 36: number analyzed (Participants) | 39
  Change at Week 36 | -34.51 (30.03)
  Change at Week 40: number analyzed (Participants) | 22
  Change at Week 40 | -34.36 (31.07)
  Change at Week 44: number analyzed (Participants) | 20
  Change at Week 44 | -32.30 (27.10)
  Change at Week 48: number analyzed (Participants) | 16
  Change at Week 48 | -35.56 (26.27)
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -36.42 (32.77)
  Change at Week 56: number analyzed (Participants) | 6
  Change at Week 56 | -39.50 (34.67)
  Change at Week 60: number analyzed (Participants) | 2
  Change at Week 60 | -42.00 (43.84)
  Change at Week 64: number analyzed (Participants) | 2
  Change at Week 64 | -40.00 (43.84)

25. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) Score at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Larger the participant's response to the questions (with the exception of 2 negatively stated questions), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). The changes from Baseline to any time point were averaged among all participants, where negative changes indicated an increase in fatigue.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 134
units on a scale
  Baseline | 25.44 (11.97)
  Change at Week 2: number analyzed (Participants) | 126
  Change at Week 2 | 3.71 (8.20)
  Change at Week 4: number analyzed (Participants) | 125
  Change at Week 4 | 6.08 (9.74)
  Change at Week 8: number analyzed (Participants) | 123
  Change at Week 8 | 7.98 (12.36)
  Change at Week 12: number analyzed (Participants) | 113
  Change at Week 12 | 9.43 (11.54)
  Change at Week 16: number analyzed (Participants) | 107
  Change at Week 16 | 9.19 (11.89)
  Change at Week 20: number analyzed (Participants) | 110
  Change at Week 20 | 8.84 (12.68)
  Change at Week 24: number analyzed (Participants) | 104
  Change at Week 24 | 9.26 (13.08)
  Change at Week 28: number analyzed (Participants) | 57
  Change at Week 28 | 11.54 (12.18)
  Change at Week 32: number analyzed (Participants) | 52
  Change at Week 32 | 9.87 (12.25)
  Change at Week 36: number analyzed (Participants) | 38
  Change at Week 36 | 8.63 (12.17)
  Change at Week 40: number analyzed (Participants) | 22
  Change at Week 40 | 10.41 (11.73)
  Change at Week 44: number analyzed (Participants) | 20
  Change at Week 44 | 10.30 (12.37)
  Change at Week 48: number analyzed (Participants) | 16
  Change at Week 48 | 11.50 (9.14)
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | 12.25 (10.70)
  Change at Week 56: number analyzed (Participants) | 6
  Change at Week 56 | 14.83 (7.36)
  Change at Week 60: number analyzed (Participants) | 2
  Change at Week 60 | 17.00 (7.07)
  Change at Week 64: number analyzed (Participants) | 2
  Change at Week 64 | 20.00 (7.07)

26. Secondary Outcome: Percentage of Participants With Health Assessment Questionnaire-Disability Index (HAQ-DI) Remission at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Description: HAQ-DI assessed 20 items in 8 functional activity domains including dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Each item was scored on a scale of 0 to 3, where 0 represented activities performed without difficulty and 3 represented inability to perform activities alone. The total score (range = 0-3) was calculated as an average of all item scores. Percentage of participants with HAQ-DI remission (HAQ-DI score <0.5) at each time point is reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 134
percentage of participants
  Baseline | 6.0
  Week 2: number analyzed (Participants) | 131
  Week 2 | 8.4
  Week 4: number analyzed (Participants) | 127
  Week 4 | 12.6
  Week 8: number analyzed (Participants) | 129
  Week 8 | 23.3
  Week 12: number analyzed (Participants) | 120
  Week 12 | 31.7
  Week 16: number analyzed (Participants) | 117
  Week 16 | 35.9
  Week 20: number analyzed (Participants) | 115
  Week 20 | 31.3
  Week 24: number analyzed (Participants) | 109
  Week 24 | 30.3
  Week 28: number analyzed (Participants) | 59
  Week 28 | 37.3
  Week 32: number analyzed (Participants) | 53
  Week 32 | 32.1
  Week 36: number analyzed (Participants) | 40
  Week 36 | 25.0
  Week 40: number analyzed (Participants) | 23
  Week 40 | 30.4
  Week 44: number analyzed (Participants) | 20
  Week 44 | 30.0
  Week 48: number analyzed (Participants) | 16
  Week 48 | 25.0
  Week 52: number analyzed (Participants) | 12
  Week 52 | 33.3
  Week 56: number analyzed (Participants) | 6
  Week 56 | 33.3
  Week 60: number analyzed (Participants) | 2
  Week 60 | 50.0
  Week 64: number analyzed (Participants) | 2
  Week 64 | 50.0

27. Secondary Outcome: Percentage of Participants With HAQ-DI Clinically Meaningful Improvement at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Description: HAQ-DI assessed 20 items in 8 functional activity domains including dressing, rising, eating, walking, hygiene, reach, grip, and usual activities. Each item was scored on a scale of 0 to 3, where 0 represented activities performed without difficulty and 3 represented inability to perform activities alone. The total score (range = 0-3) was calculated as an average of all item scores. Percentage of participants with HAQ-DI clinically meaningful improvement (reduction in HAQ-DI score from baseline >/=0.22) at each time point is reported.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, and 64
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 134
percentage of participants
  Week 2: number analyzed (Participants) | 127
  Week 2 | 42.5
  Week 4: number analyzed (Participants) | 123
  Week 4 | 55.3
  Week 8: number analyzed (Participants) | 124
  Week 8 | 62.1
  Week 12: number analyzed (Participants) | 116
  Week 12 | 71.6
  Week 16: number analyzed (Participants) | 112
  Week 16 | 75.0
  Week 20: number analyzed (Participants) | 111
  Week 20 | 67.6
  Week 24: number analyzed (Participants) | 106
  Week 24 | 73.6
  Week 28: number analyzed (Participants) | 56
  Week 28 | 76.8
  Week 32: number analyzed (Participants) | 50
  Week 32 | 72.0
  Week 36: number analyzed (Participants) | 37
  Week 36 | 64.9
  Week 40: number analyzed (Participants) | 23
  Week 40 | 73.9
  Week 44: number analyzed (Participants) | 20
  Week 44 | 65.0
  Week 48: number analyzed (Participants) | 16
  Week 48 | 62.5
  Week 52: number analyzed (Participants) | 12
  Week 52 | 50.0
  Week 56: number analyzed (Participants) | 6
  Week 56 | 66.7
  Week 60: number analyzed (Participants) | 2
  Week 60 | 100.0
  Week 64: number analyzed (Participants) | 2
  Week 64 | 50.0

28. Secondary Outcome: Treatment Compliance From Baseline up to Week 24
Description: Treatment compliance from Baseline up to Week 24 was assessed using following formula: (number of actual injection received / number of theoretical injection which should be received at week 24) * 100.
Time Frame: Baseline up to Week 24
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percentage of injections
Arm/Group | TCZ - All Participants - Core Study Period
Number analyzed (Participants) | 135
percentage of injections | 91.19 (15.54)

29. Secondary Outcome: Change From Baseline in Rheumatoid Arthritis Impact of Disease (RAID) Score at Weeks 12, 24, 28, 40, 52, and 64
Description: RAID assessed the impact of rheumatoid arthritis on participant's quality of life. It comprised 7 domains: pain, function, fatigue, physical and psychological well-being, sleep disturbance and coping. Each domain was a single question scored from 0 (best) to 10 (worst) on a continuous numerical rating scale (NRS). Each domain also had a specific weight assigned by a participant survey and RAID total score ranged from 0 (best) to 10 (worst). If only 1 domain was missing it was replaced by the mean of the others; otherwise, RAID score was not calculated. The changes from Baseline to any time point were averaged among all participants, where negative changes indicated better quality of life.
Time Frame: Baseline, Weeks 12, 24, 28, 40, 52, and 64
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 133
units on a scale
  Baseline | 5.94 (2.27)
  Change at Week 12: number analyzed (Participants) | 112
  Change at Week 12 | -2.74 (2.39)
  Change at Week 24: number analyzed (Participants) | 103
  Change at Week 24 | -2.94 (2.65)
  Change at Week 28: number analyzed (Participants) | 55
  Change at Week 28 | -2.99 (2.50)
  Change at Week 40: number analyzed (Participants) | 22
  Change at Week 40 | -3.21 (2.46)
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -3.27 (2.52)
  Change at Week 64: number analyzed (Participants) | 2
  Change at Week 64 | -5.59 (0.74)

30. Secondary Outcome: Change From Baseline in Routine Assessment of Patient Index Data 3 (RAPID-3) at Weeks 2, 4, 12, 24, 28, 40, 52, and 64
Description: RAPID-3 is a combined index derived from the Multidimensional Health Assessment Questionnaire that includes physical function score, pain VAS, and PGA VAS. The total RAPID-3 score ranges from 0 to 10 where higher scores represent worse outcomes. The changes from Baseline to any time point were averaged among all participants, where negative changes indicated better outcome.
Time Frame: Baseline, Weeks 2, 4, 12, 24, 28, 40, 52, and 64
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 134
units on a scale
  Baseline | 15.41 (6.54)
  Change at Week 2: number analyzed (Participants) | 123
  Change at Week 2 | -1.72 (4.96)
  Change at Week 4: number analyzed (Participants) | 116
  Change at Week 4 | -4.18 (6.08)
  Change at Week 12: number analyzed (Participants) | 113
  Change at Week 12 | -7.07 (7.01)
  Change at Week 24: number analyzed (Participants) | 105
  Change at Week 24 | -7.68 (7.16)
  Change at Week 28: number analyzed (Participants) | 56
  Change at Week 28 | -8.16 (6.81)
  Change at Week 40: number analyzed (Participants) | 21
  Change at Week 40 | -8.86 (6.70)
  Change at Week 52: number analyzed (Participants) | 11
  Change at Week 52 | -8.91 (7.79)
  Change at Week 64: number analyzed (Participants) | 2
  Change at Week 64 | -9.00 (9.90)

31. Secondary Outcome: Number of Participants With Patient Acceptable Symptom State (PASS) Score
Description: Participants were asked: "If you were to remain in the same condition for the next few months as you have been over the last 8 days, would this be 1) acceptable, 2) Inacceptable?" The number of participants who responded "acceptable" or "Inacceptable" at each time point is presented.
Time Frame: Baseline, Weeks 24, 52, and last assessment (up to Week 76)
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 132
Participants
  Baseline, Acceptable | 31
  Baseline, Inacceptable | 101
  Week 24, Acceptable: number analyzed (Participants) | 105
  Week 24, Acceptable | 78
  Week 24, Incceptable: number analyzed (Participants) | 105
  Week 24, Incceptable | 27
  Week 52, Acceptable: number analyzed (Participants) | 11
  Week 52, Acceptable | 8
  Week 52, Inacceptable: number analyzed (Participants) | 11
  Week 52, Inacceptable | 3
  Last Assessment, Acceptable: number analyzed (Participants) | 118
  Last Assessment, Acceptable | 83
  Last Assessment, Inacceptable: number analyzed (Participants) | 118
  Last Assessment, Inacceptable | 35

32. Secondary Outcome: Change From Baseline in Bristol Rheumatoid Arthritis Fatigue Multidimensional Questionnaire (BRAF-MDQ) Total Score at Weeks 24 and 52
Description: BRAF-MDQ assessed the overall experience and impact of disease related fatigue, using four dimensions (physical fatigue [4 items], living with fatigue [7 items], cognitive fatigue [5 items], and emotional fatigue [4 items]). A total fatigue score (range 0 to 70) was obtained by summing the 20 item scores ranging from 0 to 3, except for item 1 (0-10), item 2 (0-7) and item 3 (0-2). Higher scores reflect greater fatigue. If only 1 domain was missing it was replaced by the mean of the others; otherwise, the total score was not calculated. The changes from Baseline to any time point were averaged among all participants, where negative changes indicated better quality of life.
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 129
units on a scale
  Baseline | 35.50 (18.93)
  Change at Week 24: number analyzed (Participants) | 96
  Change at Week 24 | -13.18 (18.56)
  Change at Week 52: number analyzed (Participants) | 11
  Change at Week 52 | -20.09 (19.02)

33. Secondary Outcome: Change From Baseline in Bristol Rheumatoid Arthritis Fatigue (BRAF)-NRS Score at Weeks 24 and 52
Description: BRAF-NRS are 3 standardized NRS (range = 0-10) for disease related fatigue domains (severity of fatigue, fatigue effect, and coping with fatigue). Higher values reflect greater problems for severity/level fatigue and effect fatigue NRS, but lower scores reflect greater problems for copped fatigue NRS.
Time Frame: Baseline, Weeks 24 and 52
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 133
units on a scale
  Baseline, Level Fatigue NRS | 6.14 (2.56)
  Baseline, Effect Fatigue NRS | 5.87 (2.75)
  Baseline, Copped Fatigue NRS | 5.48 (2.52)
  Change at Week 24, Level Fatigue NRS: number analyzed (Participants) | 101
  Change at Week 24, Level Fatigue NRS | -2.41 (2.90)
  Change at Week 24, Effect Fatigue NRS: number analyzed (Participants) | 101
  Change at Week 24, Effect Fatigue NRS | -2.44 (2.90)
  Change at Week 24, Copped Fatigue NRS: number analyzed (Participants) | 101
  Change at Week 24, Copped Fatigue NRS | -0.47 (3.91)
  Change at Week 52, Level Fatigue NRS: number analyzed (Participants) | 12
  Change at Week 52, Level Fatigue NRS | -3.75 (2.93)
  Change at Week 52, Effect Fatigue NRS: number analyzed (Participants) | 12
  Change at Week 52, Effect Fatigue NRS | -3.83 (2.86)
  Change at Week 52, Copped Fatigue NRS: number analyzed (Participants) | 12
  Change at Week 52, Copped Fatigue NRS | -1.33 (2.84)

34. Secondary Outcome: Change From Baseline in Medical Outcome Study (MOS) Sleep Questionnaire Score at Weeks 12, 24, 28, 40, 52, and 64
Description: MOS sleep scale comprised of 6-item with each item score ranged from 0 to 100. The total score was the average of scores sum (range 0-100), with highest values reflecting biggest participant's sleeping problems. If more than 3 items were missing the index was not calculated. The changes from Baseline to any time point were averaged among all participants, where negative changes indicated better outcome.
Time Frame: Baseline, Weeks 12, 24, 28, 40, 52, and 64
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 133
units on a scale
  Baseline | 47.09 (21.66)
  Change at Week 12: number analyzed (Participants) | 110
  Change at Week 12 | -7.21 (18.85)
  Change at Week 24: number analyzed (Participants) | 103
  Change at Week 24 | -5.44 (19.83)
  Change at Week 28: number analyzed (Participants) | 55
  Change at Week 28 | -8.48 (15.04)
  Change at Week 40: number analyzed (Participants) | 21
  Change at Week 40 | -5.56 (14.45)
  Change at Week 52: number analyzed (Participants) | 10
  Change at Week 52 | -8.33 (18.11)
  Change at Week 64: number analyzed (Participants) | 2
  Change at Week 64 | -27.08 (2.95)

35. Secondary Outcome: Change From Baseline in Fluctuations of Disease Activity in Rheumatoid Arthritis (FLARE) Questionnaire Score at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 40, 52, and 64
Description: FLARE is a 13-item questionnaire assessed disease flares between two medical consultations. Each item score ranged from 0 (completely untrue) to 10 (absolutely true) on a 6-step scale. The FLARE questionnaire global score (range = 0-10) is a mean score of 11 of the 13 items [items 6 ('doses of pain killers or anti-inflammatory medication') and 13 ('need for help') not taken into account], with the highest score corresponding to the highest disease activity. The global score was computed if at least the scores of 6 items were available. The changes from Baseline to any time point were averaged among all participants, where negative changes indicated better outcome.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20, 24, 28, 40, 52, and 64
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 134
units on a scale
  Baseline | 5.61 (2.77)
  Change at Week 2: number analyzed (Participants) | 124
  Change at Week 2 | -1.35 (2.41)
  Change at Week 4: number analyzed (Participants) | 125
  Change at Week 4 | -2.38 (2.64)
  Change at Week 8: number analyzed (Participants) | 123
  Change at Week 8 | -2.94 (3.18)
  Change at Week 12: number analyzed (Participants) | 114
  Change at Week 12 | -3.41 (2.62)
  Change at Week 16: number analyzed (Participants) | 107
  Change at Week 16 | -3.10 (2.89)
  Change at Week 20: number analyzed (Participants) | 110
  Change at Week 20 | -3.30 (2.93)
  Change at Week 24: number analyzed (Participants) | 106
  Change at Week 24 | -3.41 (2.75)
  Change at Week 28: number analyzed (Participants) | 57
  Change at Week 28 | -3.31 (2.54)
  Change at Week 40: number analyzed (Participants) | 22
  Change at Week 40 | -3.44 (2.01)
  Change at Week 52: number analyzed (Participants) | 12
  Change at Week 52 | -4.16 (1.99)
  Change at Week 64: number analyzed (Participants) | 2
  Change at Week 64 | -7.55 (1.54)

36. Secondary Outcome: Change From Baseline in BioSecure Questionnaire Score at Week 24
Description: The BioSecure questionnaire comprised of 54-item aimed at evaluating the safety competences of participants (for example, participants' self-care safety skills and socio-demographic characteristics, type of information received, quality of life, and coping style data) treated by biologics for inflammatory arthritis and to determine the factors associated with a lower level of competences.
Time Frame: Baseline, Week 24
Population: QoL population was planned to be included in the analysis. Data for this outcome measure could not be analyzed due to unavailability of the methodology to calculate the BioSecure global score and sub-scores.
Arm/Group | TCZ - All Participants - Core Study Period
Number analyzed (Participants) | 0

37. Secondary Outcome: Percentage of Participants With Discontinuations of Corticosteroid Dosage During Core Study Period
Description: Percentage of participants with a discontinuation in corticosteroid dosage during core study period is reported. The discontinuations were categorized as either permanent or temporary. Participants with temporary discontinuation first followed by permanent discontinuation were counted in both categories. Participants who were receiving corticosteroids at Baseline were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose in core study period (overall up to 36 weeks)
Population: as for outcome 28
Measure: Number; unit: percentage of participants
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 24 | 55
percentage of participants
  Permanent Discontinuation | 8.3 | 7.3
  Temporary Discontinuation | 16.7 | 7.3

38. Secondary Outcome: Time to Permanent Discontinuation of Corticosteroid Dosage During Core Study Period
Description: Time to permanent discontinuation in corticosteroid dosage during core study period is reported. Participants who permanently discontinued corticosteroids at any time during core study period were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose in core study period (overall up to 36 weeks)
Population: as for outcome 28
Measure: Median (Full Range); unit: days
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 2 | 4
days | 24 [1 to 46] | 96 [24 to 114]

39. Secondary Outcome: Time to First Temporary Discontinuation of Corticosteroid Dosage During Core Study Period
Description: Time to first temporary discontinuation in corticosteroid dosage during core study period is reported. Participants who temporarily discontinued corticosteroids at any time during core study period were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose in core study period (overall up to 36 weeks)
Population: as for outcome 28
Measure: Median (Full Range); unit: days
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 4 | 4
days | 50 [1 to 156] | 105 [76 to 138]

40. Secondary Outcome: Percentage of Participants With Change in Corticosteroid Dosage During Core Study Period
Description: Percentage of participants with a change in corticosteroid dosage during core study period compared to Baseline is reported. The change included either an initiation/ increase (>+5mg/day prednisone or equivalent) of corticosteroid dosage or a decrease (</=-5mg/day prednisone or equivalent) of corticosteroid dosage.
Time Frame: Screening up to 8 weeks after last dose in core study period (overall up to 36 weeks)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 43 | 96
percentage of participants
  Initiation/ Increase | 0.0 | 3.1
  Decrease | 14.0 | 9.4

41. Secondary Outcome: Time to Change in Corticosteroid Dosage During Core Study Period
Description: Time to first change in corticosteroid dosage during core study period compared to Baseline is reported. The change included either an initiation/ increase (>+5mg/day prednisone or equivalent) of corticosteroid dosage or a decrease (</=-5mg/day prednisone or equivalent) of corticosteroid dosage. Participants with a change in corticosteroid dosage during core study period were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose in core study period (overall up to 36 weeks)
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for specified categories for different arms, respectively.
Measure: Median (Full Range); unit: days
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 6 | 12
days
  Initiation/ Increase: number analyzed (Participants) | 0 | 3
  Initiation/ Increase |  | 38 [23 to 50]
  Decrease: number analyzed (Participants) | 6 | 9
  Decrease | 98 [1 to 239] | 107 [25 to 225]

42. Secondary Outcome: Number of Participants According to Reasons for Change in Corticosteroid Dosage During Core Study Period
Description: Number of participants according to reasons for a change in corticosteroid dosage during core study period compared to Baseline is reported. The change included either an initiation/ increase (>+5mg/day prednisone or equivalent) of corticosteroid dosage or a decrease (</=-5mg/day prednisone or equivalent) of corticosteroid dosage. Participants with a change in corticosteroid dosage during core study period were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose in core study period (overall up to 36 weeks)
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | TCZ MONO - Core Study Period | TCZ COMBO - Core Study Period
Number analyzed (Participants) | 6 | 12
Participants
  Initiation/ Increase, Lack of Efficacy: number analyzed (Participants) | 0 | 3
  Initiation/ Increase, Lack of Efficacy | 0 | 1
  Initiation/ Increase, End of Treatment Planned: number analyzed (Participants) | 0 | 3
  Initiation/ Increase, End of Treatment Planned | 0 | 1
  Initiation/ Increase, Other Reason: number analyzed (Participants) | 0 | 3
  Initiation/ Increase, Other Reason | 0 | 1
  Decrease, Adverse Event: number analyzed (Participants) | 6 | 9
  Decrease, Adverse Event | 1 | 0
  Decrease, Lack of Efficacy: number analyzed (Participants) | 6 | 9
  Decrease, Lack of Efficacy | 0 | 1
  Decrease, End of Treatment Planned: number analyzed (Participants) | 6 | 9
  Decrease, End of Treatment Planned | 2 | 3
  Decrease, Other Reason: number analyzed (Participants) | 6 | 9
  Decrease, Other Reason | 3 | 5

43. Secondary Outcome: Percentage of Participants With Discontinuations of Corticosteroid Dosage During Study
Description: Percentage of participants with a discontinuation in corticosteroid dosage during study is reported. The discontinuations were categorized as either permanent or temporary. Participants with temporary discontinuation first followed by permanent discontinuation were counted in both categories. Participants who were receiving corticosteroids at Baseline were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose (overall up to 88 weeks)
Population: LTE population; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 40
percentage of participants
  Permanent Discontinuation | 10.0
  Temporary Discontinuation | 15.0

44. Secondary Outcome: Time to Permanent Discontinuation of Corticosteroid Dosage During Study
Description: Time to permanent discontinuation in corticosteroid dosage during study is reported. Participants who permanently discontinued corticosteroids at any time during entire study were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose (overall up to 88 weeks)
Population: as for outcome 43
Measure: Median (Full Range); unit: days
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 4
days | 202 [107 to 328]

45. Secondary Outcome: Time to First Temporary Discontinuation of Corticosteroid Dosage During Study
Description: Time to first temporary discontinuation in corticosteroid dosage during study is reported. Participants who temporarily discontinued corticosteroids at any time during entire study were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose (overall up to 88 weeks)
Population: as for outcome 43
Measure: Median (Full Range); unit: days
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 6
days | 147 [96 to 290]

46. Secondary Outcome: Percentage of Participants With Change in Corticosteroid Dosage During Study
Description: Percentage of participants with a change in corticosteroid dosage during study compared to Baseline is reported. The change included either an initiation/ increase (>+5mg/day prednisone or equivalent) of corticosteroid dosage or a decrease (</=-5mg/day prednisone or equivalent) of corticosteroid dosage.
Time Frame: Screening up to 8 weeks after last dose (overall up to 88 weeks)
Population: LTE population
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 64
percentage of participants
  Initiation/ Increase | 3.1
  Decrease | 21.9

47. Secondary Outcome: Time to Change in Corticosteroid Dosage During Study
Description: Time to first change in corticosteroid dosage during study compared to Baseline is reported. The change included either an initiation/ increase (>+5mg/day prednisone or equivalent) of corticosteroid dosage or a decrease (</=-5mg/day prednisone or equivalent) of corticosteroid dosage. Participants with a change in corticosteroid dosage during entire study were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose (overall up to 88 weeks)
Population: LTE population; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for specified categories.
Measure: Median (Full Range); unit: days
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 16
days
  Initiation/ Increase: number analyzed (Participants) | 2
  Initiation/ Increase | 44 [38 to 50]
  Decrease: number analyzed (Participants) | 14
  Decrease | 210 [96 to 428]

48. Secondary Outcome: Number of Participants According to Reasons for Change in Corticosteroid Dosage During Study
Description: Number of participants according to reasons for a change in corticosteroid dosage during study compared to Baseline is reported. The change included either an initiation/ increase (>+5mg/day prednisone or equivalent) of corticosteroid dosage or a decrease (</=-5mg/day prednisone or equivalent) of corticosteroid dosage. Participants with a change in corticosteroid dosage during entire study were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose (overall up to 88 weeks)
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 16
Participants
  Initiation/ Increase, Lack of Efficacy: number analyzed (Participants) | 2
  Initiation/ Increase, Lack of Efficacy | 1
  Initiation/ Increase, Other Reason: number analyzed (Participants) | 2
  Initiation/ Increase, Other Reason | 1
  Decrease, Lack of Efficacy: number analyzed (Participants) | 14
  Decrease, Lack of Efficacy | 1
  Decrease, End of Treatment Planned: number analyzed (Participants) | 14
  Decrease, End of Treatment Planned | 4
  Decrease, Other Reason: number analyzed (Participants) | 14
  Decrease, Other Reason | 9

49. Secondary Outcome: Number of Participants According to Reasons for Changes in csDMARDs Treatment During Core Study Period
Description: Number of participants according to reasons for changes in csDMARDs treatment during core study period is reported. The changes included Increase of dose (the dose increase had to be greater than the highest dose received within the 4 weeks on or before baseline); Addition of another csDMARD (without suppression of the first one); Switch (add and suppression) of a csDMARD for another reason than intolerance to the csDMARD suppressed; Modification of the administration route of MTX (with increase or maintenance of the dose): per oral route to intravenous (IV)/ intramuscular (IM)/ SC. Participants with a change in csDMARDs treatment during core study period were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose in core study period (overall up to 36 weeks)
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | TCZ - All Participants - Core Study Period
Number analyzed (Participants) | 29
Participants
  Adverse Event | 19
  End of Treatment Planned | 2
  Lack of Efficacy | 1
  Poor Treatment Compliance | 1
  Other Reason | 6

50. Secondary Outcome: Number of Participants According to Reasons for Changes in csDMARDs Treatment During Study
Description: Number of participants according to reasons for changes in csDMARDs treatment during study is reported. The changes included Increase of dose (the dose increase had to be greater than the highest dose received within the 4 weeks on or before baseline); Addition of another csDMARD (without suppression of the first one); Switch (add and suppression) of a csDMARD for another reason than intolerance to the csDMARD suppressed; Modification of the administration route of MTX (with increase or maintenance of the dose): per oral route to IV/IM/SC. Participants with a change in csDMARDs treatment during entire study were only included in the analysis.
Time Frame: Screening up to 8 weeks after last dose (overall up to 88 weeks)
Population: as for outcome 43
Measure: Count of Participants; unit: Participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 12
Participants
  Adverse Event | 5
  End of Treatment Planned | 1
  Lack of Efficacy | 2
  Poor Treatment Compliance | 1
  Other Reason | 3

51. Secondary Outcome: Change From Baseline in Synovitis Ultrasound B-Mode Score at Week 24
Description: Synovitis was assessed by ultrasonographic evaluation (B-mode ultrasound) and scored from "0" to "3" for each 7 paired joints (wrists on both sides, 2nd and 3rd metacarpo-phalangeal [MCP 2/3] on both sides, 2nd and 3rd proximal inter-phalangeal [PIP 2/3] on both sides, 2nd and 5th metatarsophalangeal [MTP 2/5] on both sides). Synovitis total score was calculated by adding the sum of scores for each joint for a total score ranging from 0 to 42. A score of 0 indicated no damage and a score of 42 indicated most severe damage. The changes from Baseline to any time point were averaged among all participants, where negative changes indicated better outcome.
Time Frame: Baseline, Weeks 24
Population: FAS; Here, 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies number of participants evaluable for specified categories.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 74
units on a scale
  Baseline | 14.0 [2.0 to 37.0]
  Change at Week 24: number analyzed (Participants) | 54
  Change at Week 24 | -8.0 [-29.0 to 8.0]

52. Secondary Outcome: Change From Baseline in Synovitis Ultrasound Power-Doppler Mode Score at Week 24
Description: Synovitis was assessed by ultrasonographic evaluation (Power-Doppler-mode ultrasound) and scored from "0" to "3" for each 7 paired joints (wrists on both sides, 2nd and 3rd metacarpo-phalangeal [MCP 2/3] on both sides, 2nd and 3rd proximal inter-phalangeal [PIP 2/3] on both sides, 2nd and 5th metatarsophalangeal [MTP 2/5] on both sides). Synovitis total score was calculated by adding the sum of scores for each joint for a total score ranging from 0 to 42. A score of 0 indicated no damage and a score of 42 indicated most severe damage. The changes from Baseline to any time point were averaged among all participants, where negative changes indicated better outcome.
Time Frame: Baseline, Weeks 24
Population: as for outcome 51
Measure: Median (Full Range); unit: units on a scale
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 74
units on a scale
  Baseline | 5.0 [0.0 to 26.0]
  Change at Week 24: number analyzed (Participants) | 54
  Change at Week 24 | -4.0 [-21.0 to 11.0]

53. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies to Tocilizumab
Description: Percentage of participants with a positive response to anti-therapeutic antibodies against tocilizumab by confirmatory assays at any time during the study is reported.
Time Frame: Baseline up to 8 weeks after last study drug administration (up to Week 84)
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | TCZ - All Participants
Number analyzed (Participants) | 139
percentage of participants | 3.6

ADVERSE EVENTS:
Time Frame: Baseline up to 8 weeks after last study drug administration (up to Week 84)
Description: Treatment-emergent adverse events (TEAEs) are adverse events occurring between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. FAS.
Groups:
- TCZ MONO - All Participants: Participants who did not receive treatment with any csDMARDs 4 weeks prior first TCZ administration and received monotherapy with TCZ at a dose of 162 mg as SC injection once a week for 24 weeks. Participants who completed the core study period were allowed to enter a LTE period to continue study treatment for up to a maximum of another 52 weeks or until the commercial availability of SC TCZ, whichever came first.
- TCZ COMBO - All Participants: Participants who received treatment with MTX or other csDMARDs 4 weeks prior first TCZ administration and/or received TCZ at a dose of 162 mg as SC injection once a week in combination with MTX or other csDMARDs (at investigator's discretion) for 24 weeks. Participants who completed the core study period were allowed to enter a LTE period to continue study treatment for up to a maximum of another 52 weeks or until the commercial availability of SC TCZ, whichever came first.
Arm/Group | TCZ MONO - All Participants | TCZ COMBO - All Participants | TCZ - All Participants
Serious Adverse Events (participants affected / at risk) | 5/43 | 11/96 | 16/139
Other Adverse Events (participants affected / at risk) | 28/43 | 65/96 | 93/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TCZ MONO - All Participants (N=43) | TCZ COMBO - All Participants (N=96) | TCZ - All Participants (N=139)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 1
Gastric volvulus (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Disseminated tuberculosis (Infections and infestations) | 0 | 1 | 1
Meningitis tuberculous (Infections and infestations) | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TCZ MONO - All Participants (N=43) | TCZ COMBO - All Participants (N=96) | TCZ - All Participants (N=139)
Bronchitis (Infections and infestations) | 7 | 9 | 16
Ear infection (Infections and infestations) | 5 | 3 | 8
Nasopharyngitis (Infections and infestations) | 4 | 8 | 12
Rhinitis (Infections and infestations) | 2 | 11 | 13
Urinary tract infection (Infections and infestations) | 4 | 4 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 8 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 9
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 8 | 11 | 19
Abdominal pain (Gastrointestinal disorders) | 0 | 5 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 9
Nausea (Gastrointestinal disorders) | 4 | 2 | 6
Asthenia (General disorders) | 1 | 9 | 10
Injection site erythema (General disorders) | 4 | 3 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 6
Psoriasis (Skin and subcutaneous tissue disorders) | 4 | 0 | 4
Alanine aminotransferase increased (Investigations) | 2 | 8 | 10
Transaminases increased (Investigations) | 0 | 5 | 5
Headache (Nervous system disorders) | 2 | 8 | 10
Neutropenia (Blood and lymphatic system disorders) | 2 | 7 | 9
Hypertension (Vascular disorders) | 3 | 2 | 5
Insomnia (Psychiatric disorders) | 0 | 5 | 5
Hepatocellular injury (Hepatobiliary disorders) | 1 | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.